CLINICAL TRIAL: NCT06243120
Title: Intravenous Lidocaine for Treating Intrathecal Fentanyl Induced Pruritus
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Sabah Nageeb, Lecturer of anesthesia, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KACS, KSA: H-08- L-074
Record Dates: First submitted 2024-01-19; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-01

CONDITIONS: Pruritus Caused by Drug
Keywords: Spinal anesthesia; Pruritus; Lidocaine
MeSH Terms: conditions — Pruritus

STUDY DESIGN:
Intervention Model Description: Randomized, prospective trial on 2 equal groups
Who Masked: Care Provider
Masking Description: Preparation of the used infusion volume will performed by anesthesia specialist in our center not sharing in the study, he is the one who know it is placebo or lidocaine. The infusion performed blindly by the researcher and VAS will be assessed by the circulating nurse inside the theater or the nurse in the PACU.
  The regression of VAS in comparison to initial pruritus scale will be recorded in both groups. The percentage of incidence of pruritus, body distribution of pruritus, duration of spinal anesthesia and local anesthetic toxicity symptoms will be recorded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): The study group will receive lidocaine (2%) 1mg/ kg iv diluted by normal saline to a volume of 100 ml. The VAS will be assessed every 10 minutes for 60minutes after the treatment. A regression of more than 4 points of VAS score is considered a success and if less than 4 points, it is considered as a failure.
  If intravenous lidocaine failed to manage pruritus after 30 minutes the patient will receive 20 mg intravenous propofol.
  Interventions: Drug: Lidocaine IV
- Control group (Placebo Comparator): The control group will receive 100 ml of normal saline as placebo effect and VAS will be assessed every 10 minutes for 60minutes after the treatment. A regression of more than 4 points of VAS score is considered a success and if less than 4 points, it is considered as a failure.
  If intravenous lidocaine failed to manage pruritus after 30 minutes the patient will receive 20 mg intravenous propofol.
  Interventions: Drug: Lidocaine IV

INTERVENTIONS:
Drug: Lidocaine IV — The study group will receive lidocaine (2%) 1mg/ kg iv diluted by normal saline to a volume of 100 ml. The VAS will be assessed every 10 minutes for 60minutes after the treatment. A regression of more than 4 points of VAS score is considered a success and if less than 4 points , it will be considered as a failure.

SUMMARY:
The study will assess efficacy of intravenous lidocaine 1 mg/kg diluted with 0.9% sodium chloride to a volume of 100 ml to suppress intrathecal fentanyl induced pruritus. This will be compared to control group who will receive 100 ml normal saline as placebo.

The main outcome is regression of initial VAS score with incidence of pruritus.

DETAILED DESCRIPTION:
The study will include adult patients who are admitted for orthopedic operations and Urosurgery who are planned to receive spinal anesthesia. The study will include adult patients aging from 18 to 70 years old. ASA I to III. The study will exclude the patients who receive antihistamine drugs, patients who suffer any type of coagulopathy, patients who are suffering any type of pruritus before receiving spinal anesthesia and patients who are known allergic to lidocaine. All the patients will receive 500 ml ringer lactate as a volume preload. The patients will be monitored by SPO2, Noninvasive blood pressure and ECG. The spinal anesthesia drugs will be hyperbaric bupivacaine (the dose will be adjusted according to the required level of anesthesia) and 25 mic of fentanyl as an additive. The subjects of the study will not receive any type of sedation. If any patient suffered bradycardia associated with hypotension which necessitate management by atropine or ephedrine, he will be excluded from the study.

Before the surgery, patients could cooperate and understand the Visual Analogue Score (VAS) scale. Patients will be explained about the use of VAS for grading the severity of pruritus on a scale of 0 to 10. VAS = 0 means no pain or itching, VAS = 10 means worst sensation and VAS > 4 means it need intervention. The affected areas by itching will be asked.

The study group will receive lidocaine (2%) 1mg/ kg iv diluted by normal saline to a volume of 100 ml. The VAS will be assessed every 10 minutes for 60minutes after the treatment. A regression of more than 4 points of VAS score is considered a success and if less than 4 points , it will be considered as a failure.

The control group will receive 100 ml of normal saline as placebo effect and VAS will be assessed in same manner as the study group.

ELIGIBILITY:
Inclusion Criteria:

* patients who are admitted for orthopedic operations and Urosurgery who are planned to receive spinal anesthesia.
* The study will include adult patients aging from 18 to 70 years old. ASA I to III.

Exclusion Criteria:

* the patients who receive antihistamine drugs
* patients who suffer any type of coagulopathy
* patients who are suffering any type of pruritus before receiving spinal anesthesia
* patients who are known allergic to lidocaine.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
regression of VAS in comparison to initial pruritus scale. | The whole perioperative period
  Before the surgery, patients could cooperate and understand the Visual Analogue Score (VAS) scale. The patients will be explained about the use of VAS for grading the severity of pruritus on a scale of 0 to 10. VAS = 0 means no pain or itching, VAS = 10 means worst sensation and VAS > 4 means it needs intervention.

SECONDARY OUTCOMES:
The percentage of incidence of pruritus | The whole perioperative period
  observation
body distribution of pruritus | The whole perioperative period
  observation
local anesthetic toxicity symptoms. | The whole perioperative period
  observation

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Through the official email

REFERENCES:
- [Background] Wang J, Li J, Cao H, Zhou X, Tang Q. Intravenous lidocaine suppresses dexamethasone-induced perineal pruritus during anesthesia induction: a randomized controlled, double blind study. Pak J Pharm Sci. 2015 Mar;28(2):569-72. PMID 25730811